CLINICAL TRIAL: NCT05498441
Title: Neuroimaging Biomarker-guided Personalized High-Definition Transcranial Direct Current Stimulation (HD-tDCS) Treatment for Major Depressive Episode in Adolescents With Mood Disorders: A Randomized Controlled Study
Brief Title: Personalized High-Definition Transcranial Direct Current Stimulation (HD-tDCS) Treatment for Major Depressive Episode
Acronym: PRHDTDCSTMDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81725005-3
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Major Depressive Episode
Keywords: High-Definition Transcranial Direct Current Stimulation; Major Depressive Episode; Magnetic Resonance Imaging; Adolescent
MeSH Terms: interventions — Antipsychotic Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized HD-tDCS (Experimental): The experimental arm will receive the personalized HD-tDCS treatment with parameters as follows:
  1. Neuroimaging biomarker-guided personalized selection for central electrode polarity: anode or cathodal;
  2. Neuroimaging biomarker-guided personalized selection for stimulation site: dorsalmedial prefrontal cortex or occipital cortex;
  3. Schedule: 2 sessions per day, five days per week for a total of 20 sessions over 2 weeks.
  Interventions: Device: High-Definition Transcranial Direct Current Stimulation (HD-tDCS); Drug: Antipsychotics, mood stabilizers, etc.
- Routine HD-tDCS (Active Comparator): Routine stimulation arm will receive the same scheme of HD-tDCS, but the stimulation target is L-DLPFC with anode as central electrode.
  Interventions: Device: High-Definition Transcranial Direct Current Stimulation (HD-tDCS); Drug: Antipsychotics, mood stabilizers, etc.

INTERVENTIONS:
Device: High-Definition Transcranial Direct Current Stimulation (HD-tDCS) — High-Definition Transcranial Direct Current Stimulation (HD-tDCS) is a non-invasive neuromodulation therapy which has been recognized as a helpful treatment for depression. During each HD-tDCS treatment, the electrode field is generated by a 4*1 ring montage which is placed over the scalp on the brain region of interest with an electrical current induced to modulate brain activity.
Drug: Antipsychotics, mood stabilizers, etc. — During the HD-tDCS treatment period, all the participants will maintain the stable medication regimen according to clinical practice guidelines.

SUMMARY:
Adolescents with mood disorders experiencing major depressive episode have poor efficacy of medication treatment. High-Definition Transcranial Direct Current Stimulation (HD-tDCS) has been proven adjuvant efficacy in patients with major depressive episode. However, the optimal evidence-based stimulation parameters have not been clearly defined, which greatly limits the efficacy of HD-tDCS in the treatment of major depressive episode.This trial will compare a novel form of accurate and personalized HD-tDCS treatment protocol guided by neuroimaging biomarkers to the routine stimulation(stimulation target is L-DLPFC, central electrode is anode).The personalized selection of stimulation site, central electrode polarity will be determined by neuroimaging biomarkers. The study aims to propose a novel personalized neuroimaging-guided HD-tDCS strategy, to evaluate the efficacy and safety of the treatment, further to understand the biological mechanism of the personalized HD-tDCS treatment.

DETAILED DESCRIPTION:
Mood disorders, including mainly bipolar disorder (BD) and major depressive disorder (MDD), have become the primary health problem and one of the leading causes of functional disability in adolescents . In China, the incidence of mood disorders such as BD and MDD in adolescence has increased rapidly in recent years. Particularly, patients with mood disorder currently experiencing major depressive episode have high risk of suicide, and pharmacological treatment showed poor efficacy to such depressive patients. Mood disorders with major depressive episode have become one of the major threats to the mental health of adolescents in China. Therefore, it is of great significance to explore a series of early intervention strategies for adolescents with major depressive episode. HD-tDCS is a non-invasive brain stimulation treatment strategy with mild side effects. The set of stimulation parameters often has a vital impact on the final clinical efficacy of HD-tDCS treatment. Several clinical trials have reported the efficacy and safety of HD-tDCS on treatment major depression disorder. However, the evidence-based optimal targets and other stimulation parameters have not been clearly defined, which greatly limits the efficacy of HD-tDCS in the treatment of major depressive episode. To date, there is no large randomized clinical trial (RCT) exploring an optimization of HD-tDCS on adolescents with major depressive episode. This study is a randomized controlled trial aiming at assessing the efficacy and safety of a novel personalized HD-tDCS treatment protocol compared to routine stimulation for major depressive episode in adolescents with mood disorders. Participants will be assigned randomly (1:1) to the personalized HD-tDCS group or the routine HD-tDCS group. Participants will be treated with 20 sessions (2 sessions per day) HD-tDCS treatment. The stimulation parameters of routine HD-tDCS group are: current=2 mA, duration=20 min, stimulation target=L-DLPFC, central electrode=anode. The stimulation parameters of personalized HD-tDCS group are current=2 mA and duration=20 min, while the stimulation target and central electrode polarity are based on neuroimaging biomarkers extracted via machine learning. Participants in both groups will maintain the stable drug regimen during the HD-tDCS trial.

ELIGIBILITY:
Inclusion Criteria:

* Between 13 and 18 years of age;
* Participants fulfill the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnostic criteria for major depressive disorder (MDD) or bipolar disorder (BD);
* Participants are assessed by the Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime version (K-SADS-PL);
* A current moderate or severe depressive episode defined by HAMD>17;
* Participants receive a stable psychotropic medication regimen prior to randomization to the trial and patient will be willing to remain on the stable regimen during the HD-tDCS treatment phase;
* All participants provided written informed consent by themselves or their guardians after the detailed description of the study.

Exclusion Criteria:

* Prior rTMS, tDCS, electroconvulsive therapy (ECT) application or standard psychological therapy within 6 months prior to screening;
* Comorbidity of other DSM-IV axis I disorders or personality disorders;
* Judged clinically to be at serious suicidal risk;
* Diabetes mellitus, hypertension, vascular and infectious diseases and other major medical comorbidities;
* Unstable medical conditions, e.g., severe asthma;
* Neurological disorders, e.g., history of head injury with loss of consciousness for ≥ five minutes, cerebrovascular diseases, brain tumors and neurodegenerative diseases;
* Mental retardation or autism spectrum disorder;Contraindications to MRI (e.g., severe claustrophobia, pacemakers, metalimplants);
* Contraindications to HD-tDCS (e.g., scalp rupture, cranial plates, history of seizure,electroencephalogram (EEG) test suggesting high risk of seizure, known brain lesion);
* Current drug/alcohol abuse or dependence;Pregnant or lactating female.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms assessed by Hamilton depression rating scale 17 items (HAMD-17) at week 1 and week 2. | Baseline, week 1 and week 2
  The HAMD-17 scale has 17 items. The total score ranges from 0-52, with higher score indicating more severe depressive symptoms. A total score of 0-7 is considered to be normal. Scores of 17 or higher indicate moderate, severe, or very severe depression.
Change from baseline in neurocognitive function using Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) test at week 2. | Baseline and week 2.
  RBANS is a test for identifying and characterizing abnormal cognitive decline for patients with neuropsychiatric disorders. The RBANS is comprised of five domains, which are Immediate Memory, Visuospatial /Constructional,Language, Attention and Delayed Memory. The total score of RBANS range from 40-160, with 160 referring to higher cognitive functioning. A score of 95-115 is in the average range; score of 70-85 mild to moderate cognitive impairment; score <70 moderate to severe impairment.
Change from baseline in resting-state magnetic resonance imaging (MRI) , diffusion tensor imaging (DTI) and structural (T1-weighted) imaging at weeks 1 and 2. | Baseline, week 1 and week 2.
  Participants will undergo MRI scans prior to beginning HD-tDCS treatment (week 0) and after completing 10 sessions of HD-tDCS treatment (weeks 1) and after completing 20 sessions of HD-tDCS treatment (weeks 2). This allows for a comprehensive examination of changes from baseline in functional activity, DTI and structural changes in the brain at weeks 1 and 2.

SECONDARY OUTCOMES:
Change from baseline in the Clinical Global Impression-Severity scale (CGI-S) at week 1 and week 2. | Baseline, week 1 and week 2.
  The CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. A rating of 1 is considered normal, or with the least severe symptoms, a rating of 7 is extremely ill, or the worst symptoms.
Change from baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) at week 1 and week 2. | Baseline, week 1 and week 2.
  MADRS is a clinician-rated scale used to assess depressive symptom severity and detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is rated from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms). The total score of MADRS ranges from 0 to 60, with higher score indicating more severe depression.
Change from baseline in depressive symptoms assessed by the Patient Health Questionnaire-9 (PHQ-9; range: 0-27) at baseline, week 1 and week 2. | Baseline, week 1 and week 2.
  The total scores of these questionnaires were interpreted as follows: normal (0-4), mild (5-9), moderate (10-14), and severe (15-27) depression.
Change from baseline in anxiety symptoms assessed by the Generalized Anxiety Disorder-7 (GAD-7, range: 0-21) at baseline, week 1 and week 2. | Baseline, week 1 and week 2.
  The total scores of these questionnaires were interpreted as follows: normal (0-4), mild (5-9), moderate (10-14), and severe (15-21) anxiety.
Change from baseline in insomnia symptoms assessed by the Insomnia Severity Index (ISI; range: 0-28) at baseline, week 1 and week 2. | Baseline, week 1 and week 2.
  The total scores of these questionnaires were interpreted as follows: normal (0-7), mild (8-14), moderate (15-21), and severe (22-28) insomnia.
Change from baseline in suicidal ideation assessed by the Beck Scale for Suicide (BSS-14; range: 0-38) at baseline, week 1 and week 2. | Baseline, week 1 and week 2.
  The total scores of these questionnaires were interpreted as follows: no or low suicidal ideation (0-8), moderate suicidal ideation (9-16), high suicidal ideation (17-38).
Change from baseline in perceived stress assessed by the Perceived Stress Scale-14 (PSS-14; range: 0-56) at baseline, week 1 and week 2. | Baseline, week 1 and week 2.
  The total scores of these questionnaires were interpreted as follows: normal (0-28), moderate (29-42), severe (43-56).
Change from baseline in neurocognitive function using Wsiconsin card sorting test (WCST) at week 2. | Baseline and week 2.
  The Wisconsin Card Sorting Test measures the ability to categorize, generalize, working memory, and cognitive transfer based on previous experience. Cognitive functions reflected include: abstract generalization, cognitive transfer, attention, working memory, information extraction, categorization maintenance, categorization switching, stimulus reconsideration and processing, sensory input, and motor output.
Change from baseline in neurocognitive function using Verbal Emotion Perception Test (VEPT) at week 2. | Baseline and week 2.
  VEPT can be used to identify the patient's ability to perceive emotions contained in speech, including the seven emotions of calmness, anger, sadness, fear, surprise, sarcasm, and disgust.
Change from baseline in neurocognitive function using Facial Emotion Perception Test (FEPT) at week 2. | Baseline and week 2.
  The FEPT can be used to recognize a patient's ability to perceive the emotions contained in a face, including the seven emotions of calmness, anger, disgust, fear, happiness, sadness, and surprise.
Change from baseline in acoustic features. | Baseline, week 1 and week 2.
  Participants will record videos prior to beginning intervention (baseline) and after completing intervention (week 1, week 2). Acoustic features (Hz) are a set of indicators that can reflect an individual's emotional state.
Change from baseline in manic symptoms assessed by the Young Manic Rating Scale(YMRS) at baseline, week 1 and week 2. scales. | Baseline, week 1 and week 2.
  The total scores of these questionnaires were interpreted as follows: normal (0-5), mild (6-12), moderate (13-19), and severe (20-29) manic.
Changes from metabolites in peripheral blood. | Baseline, week 1 and week 2.
  Peripheral blood samples were collected from all participants at baseline, week 1 and week 2. Plasma samples were obtained and stored at -80°C. We will conducted untargeted metabolomics analysis to obtained metabolomic data. Metabolomics is the scientific study of chemical processes involving metabolites, the small molecule substrates, intermediates, and products of cell metabolism.
Changes from protein samples in peripheral blood. | Baseline, week 1 and week 2.
  Peripheral blood samples were collected from all participants at baseline, week 1 and week 2. Data Independent Acquisition (DIA) mass spectrometry methods were employed to acquire and analyze protein samples. High- and low-abundance proteins are collected and digested into peptides using the Agilent Multiple Affinity Removal System and Filter-Assisted Sample Preparation (FASP). Data dependent acquisition (DDA) mass spectrometry analysis was then performed by Q-Exactive HF-X mass spectrometry to generate DDA libraries.
Changes from methylation in peripheral blood. | Baseline, week 1 and week 2.
  Peripheral blood samples were collected from all participants at baseline, week 1 and week 2. Epigenetics data were obtained by processing DNA samples and hybridizing them to the Illumina Infinium Methylation EPIC BeadChip, which enables quantitative assessment of over 850,000 methylation sites across the genome at single-nucleotide resolution, following the Infinium HD Methylation Assay Protocol.
Electroencephalogram - delta waves (0.5-4 Hz) | Baseline
  We collecte brainwave frequencies including delta waves (0.5-4 Hz), theta waves (4-8 Hz), alpha waves (8-13 Hz), beta waves (13-30 Hz), and gamma waves (above 30 Hz).
  Delta Waves (0.5-4 Hz) are typically recorded during deep sleep. EEG recordings are made using electrodes placed on the scalp while the person is sleeping, preferably during non-REM (rapid eye movement) sleep stages.
Electroencephalogram - theta waves (4-8 Hz) | Baseline
  We collecte brainwave frequencies including delta waves (0.5-4 Hz), theta waves (4-8 Hz), alpha waves (8-13 Hz), beta waves (13-30 Hz), and gamma waves (above 30 Hz).
  Theta Waves (4-8 Hz) are commonly observed during light sleep and the early stages of sleep. EEG recordings are made in a similar way to delta waves, during sleep stages where theta activity is predominant.
Electroencephalogram - alpha waves (8-13 Hz) | Baseline
  We collecte brainwave frequencies including delta waves (0.5-4 Hz), theta waves (4-8 Hz), alpha waves (8-13 Hz), beta waves (13-30 Hz), and gamma waves (above 30 Hz).
  Alpha Waves (8-13 Hz) are most prominent when a person is awake but relaxed, with eyes closed. EEG electrodes are placed on the scalp during a relaxed state, such as during meditation or when a person is awake but resting.
Electroencephalogram - Beta Waves (13-30 Hz) | Baseline
  We collecte brainwave frequencies including delta waves (0.5-4 Hz), theta waves (4-8 Hz), alpha waves (8-13 Hz), beta waves (13-30 Hz), and gamma waves (above 30 Hz).
  Beta Waves (13-30 Hz)are observed when a person is awake and engaged in mental activities, such as problem-solving or active thinking. EEG recordings are made during tasks that require concentration and mental effort.
Electroencephalogram- gamma waves (above 30 Hz) | Baseline
  We collecte brainwave frequencies including delta waves (0.5-4 Hz), theta waves (4-8 Hz), alpha waves (8-13 Hz), beta waves (13-30 Hz), and gamma waves (above 30 Hz).
  Gamma Waves (Above 30 Hz) are the fastest documented brain wave activity and are often associated with higher mental activities such as perception and consciousness. They are recorded using advanced EEG techniques and are typically observed during complex cognitive tasks.
Change from baseline in psychotic symptoms assessed by the Brief Psychiatric Rating Scale (BPRS) at baseline, week 1 and week 2. scales. | Baseline, week 1 and week 2.
  The total scores of these questionnaires were interpreted as follows: normal (0-35) and abnormal (>35) .
Change from baseline in anxious symptoms assessed by the Hamilton anxiely scale (HAMA) at baseline, week 1 and week 2. scales. | Baseline, week 1 and week 2.
  The total scores of these questionnaires were interpreted as follows: normal (0-7), mild (8-14), moderate (15-21), and severe (22-28) manic.
Change from baseline in anhedonia symptoms assessed by the Snaith-Hamilton Pleasure Scale(SHAPS) at baseline, week 1 and week 2. | Baseline, week 1 and week 2.
  The total scores of these questionnaires were interpreted as follows: normal (0-7) and abnormal (>7) .
Change from baseline in anhedonia symptoms assessed by the Temporal Experience of Pleasure Scale (TEPS) at baseline, week 1 and week 2. | Baseline, week 1 and week 2.
  The scale consists of two subscales: Anticipatory Pleasure and Consummatory Pleasure, each containing 18 items. The total scores for Anticipatory Pleasure and Consummatory Pleasure range from 0 to 54, with higher scores indicating a richer experience of pleasure. Generally, higher total scores are considered meaningful, while lower scores may indicate a decrease or lack of pleasure experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Wang, Study Chair — Affiliated Nanjing Brain Hospital, Nanjing Medical University
Locations (1):
- Affiliated Nanjing Brain Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No